CLINICAL TRIAL: NCT03085485
Title: A Randomized, Double-blind, Phase 2, Placebo Controlled Study to Determine the Safety and Efficacy of Ivacaftor (VX-770) for the Treatment of Chronic Obstructive Pulmonary Disease (The Topic Trial)
Brief Title: The Topic Trial - Study to Determine the Safety and Efficacy of Ivacaftor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Principal Investigator, Mark Dransfield, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F160920009; 1R34HL127166-01 (NIH)
Record Dates: First submitted 2017-02-16; First posted 2017-03-21 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Bronchitis
Keywords: COPD; CFTR; ivacaftor; topic trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — ivacaftor

STUDY DESIGN:
Intervention Model Description: The design is a pilot, randomized (3:1, active:placebo), double-blind, placebo-controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ivacaftor (Active Comparator): Ivacaftor, 150 mg PO every 12 hrs for 84 days
  Interventions: Drug: Ivacaftor 150 MG
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivacaftor 150 MG — Ivacaftor is a CFTR potentiator
  Other Names: KALYDECO
  Arms: Ivacaftor
Drug: Placebo — placebo pills
  Arms: Placebo

SUMMARY:
The study is a Phase 2 Study to establish the safety and efficacy of a drug called Ivacaftor (VX-770) in patients with chronic obstructive pulmonary disease (COPD), chronic bronchitis, and acquired CFTR dysfunction as detected by sweat chloride analysis. The design is a pilot, randomized (3:1, active:placebo), double-blind, placebo-controlled study. Approximately 40 subjects with COPD will be randomized.

DETAILED DESCRIPTION:
Like CF, COPD is characterized by small airway mucus obstruction that is associated with accelerated loss of lung function and mortality. Preliminary data indicate that cigarette smoke exerts deleterious effects on airway epithelial function including the reduction of CFTR activity, enhanced mucus expression, and a pronounced reduction in mucociliary transport (MCT). Preliminary data also indicate that approximately 50% of patients with COPD have reduced CFTR activity, as detected in the upper airways, lower airways and sweat glands. Furthermore, CFTR dysfunction is independently associated with chronic bronchitis, can persist despite smoking cessation, and can be reversed by the CFTR potentiator ivacaftor (VX-770) in vitro by activating wild-type CFTR, resulting in a robust increase in MCT. Combined with unprecedented clinical improvement via augmented mucociliary clearance in CF patients with a responsive CFTR mutation treated with ivacaftor, these data indicate that CFTR represents a viable therapeutic target to address mucus stasis in a large subset of COPD patients (potentially representing over 4 million patients in the U.S. alone). This project will investigate the hypothesis that ivacaftor can augment CFTR activity in individuals with COPD who exhibit chronic bronchitis, resulting in meaningful improvements in epithelial function and respiratory health. The investigators' initial pilot study in patients with COPD and chronic bronchitis demonstrated that ivacaftor was safe, demonstrated stable pharmacokinetics, and exhibited a trend towards efficacy in measures of PROs and sweat chloride. The current trial will test the safety, pharmacokinetics, and pharmacodynamics of ivacaftor in a larger number of COPD patients with chronic bronchitis and for a longer treatment period, evaluating the potential of CFTR potentiator therapy to address acquired CFTR dysfunction in this population and set the stage for larger and longer-term trials in the future. Based on an IND already in place in the Rowe laboratory, an IRB familiar with the proposed study, an experienced clinical investigation team with expertise in all of the endpoints proposed, and a well characterized COPD population prioritized for the presence chronic bronchitis, CFTR dysfunction, and the absence of congenital CFTR mutations, the investigators are poised to deliver the trial.

Enrollment is planned at a single center, The University of Alabama at Birmingham. Patients will be randomized 3:1 to active drug (n=30) and placebo (10) to achieve the enrollment goal.

A sufficient number of subjects will be screened to randomize up to 50 subjects to achieve 40 completed subjects to receive either ivacaftor 150 mg BID (n=30) or placebo (n=10) for 84 days.

Ivacaftor and matching placebo will be orally administered as capsules according to the following guidelines:

Between study visit Day 1 and study visit Day 84, subjects will take 1 dose of study drug each day in the morning, beginning any time between 08:00 h (8:00 AM) and 12:00 h (12:00 PM). Whenever possible, subjects should take the study drug at the same time each day.

On the study visit days when PK samples are collected (study visit Days 1, 28, 56, and 84), the study drug is to be taken by the subject while he/she is at the study site

For visits after the Day 1 visit, subjects will be instructed to bring all remaining study drug materials to the site; study drug will be dispensed at each visit.

Ivacaftor will be prepared and dispensed by an unblinded pharmacist.

Subjects will be instructed to continue their standard COPD medication regimen.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 40-80
* A Clinical diagnosis of COPD as defined by GOLD
* At Least a 10 pack year smoking history
* Exhibit symptoms of chronic bronchitis as defined by the Medical Research Council
* FEV1% predicted ≥ 35% and ≤70% Post Bronchodilator
* Clinically stable in the last 4 weeks with no evidence of COPD exacerbation
* Weight of 40 kg-120 kg
* Willingness to use at least one form of acceptable birth control including abstinence, condom with spermicide, or hormonal contraceptives from time of signing ICF through study follow up visit
* Willing to monitor blood glucose if known history of diabetes mellitus requiring insulin or medical therapy
* Element of CFTR Dysfunction, as defined by Sweat Chloride > 30 mEq/L)

Exclusion Criteria:

* Current Diagnosis of Asthma
* Known Diagnosis of Cystic Fibrosis
* Use of Continuous Oxygen Therapy of greater than 2 liters per minute - patients on 2 liters of Oxygen or less will be excluded if they have been hospitalized for COPD in the prior year or had more than 2 exacerbations requiring steroids and/or antibiotics in the prior year.
* Documented history of drug abuse within the last year
* Subjects should not have a pulmonary exacerbation or changes in therapy for pulmonary disease within 28 days before receiving the first dose of study drug.
* Cirrhosis or elevated liver transaminases > 3X ULN
* GFR < 50 estimated by Cockroft-Gault
* Any illness or abnormal lab finding that, in the opinion of the investigator might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Pregnant or Breastfeeding
* Subjects taking moderate or strong inhibitors or inducers of CYP3A4, including certain herbal medications and grapefruit juice. (Excluded medications and foods including the drugs and foods listed in the IRB HSP application.)
* Uncontrolled Diabetes
* Recent (e.g 1year) arterial thrombotic events (peripheral arterial disease, thrombotic stroke)
* Clinically significant arrhythmias requiring anti-arrhythmic agent(s) or conduction abnormalities that in the opinion of the investigator that affect patient safety such as the abnormalities listed below (patients with stable coronary artery disease are eligible) : (1) Angina symptoms (2) History of MI (3) Revascularization procedure in the last year prior to screening (4) Clinically significant congestive heart failure (known LVEF <= 45%, cor pulmonale, diastolic heart failure, etc)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Lung Health Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vijaykumar K, Solomon GM, Guimbellot J, Acosta EP, Bhambhavni PG, White S, Kim H, Raju SV, Rasmussen LW, Harris N, Liu B, Hathorne H, Rowe SM, Dransfield MT. Ivacaftor for Chronic Obstructive Pulmonary Disease: Results from a Phase 2, Randomized Controlled Trial. Am J Respir Crit Care Med. 2025 May;211(5):823-831. doi: 10.1164/rccm.202407-1302OC. PMID 39316773

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ivacaftor | Placebo
Started | 30 | 10
Completed | 28 | 10
Not Completed | 2 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ivacaftor: Ivacaftor, 150 mg PO BID for 84 days
  Ivacaftor 150 MG: Ivacaftor is a CFTR potentiator
- Total: Total of all reporting groups
Arm/Group | Ivacaftor | Placebo | Total
Number analyzed (Participants) | 30 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (7.9) | 65.9 (5.3) | 65.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 19 | 4 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 4 | 15
  White | 19 | 6 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (5.7) | 28.0 (5.3) | 27.7 (5.6)
Current Smoker [Count of Participants; unit: Participants] | 20 | 4 | 24
Smoking Exposure [Mean (Standard Deviation); unit: pack/year] | 41.3 (25.2) | 27.8 (15.4) | 38.0 (22.7)

OUTCOME MEASURES:

1. Primary Outcome: Safety of Ivacaftor - Number of Participants With Adverse Events
Description: Safety of ivacaftor will be determined by number of participants with adverse events (including serious adverse events).
Time Frame: From Screening to Day 98
Population: One subject dropped out of study after being randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 29 | 10
Participants
  Subject with any AE | 19 | 6
  AE resulting in drug interruption | 7 | 3
  AE resulting in drug discontinuation | 1 | 1

2. Primary Outcome: Safety of Ivacaftor - Number of Participants With Abnormal Serum Chemistry
Description: Number of participants with abnormal serum chemistry values compared to screening values will also be used to determine safety of ivacaftor.
Time Frame: From Screening to Day 98
Measure: Count of Participants; unit: Participants
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 29 | 10
Participants | 0 | 0

3. Primary Outcome: Safety of Ivacaftor - Number of Participants With Abnormal Hematology
Description: Safety of ivacaftor will also be determined by number of participants with abnormal changes in their screening hematology values.
Time Frame: From Screening to Day 98
Measure: Count of Participants; unit: Participants
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 29 | 10
Participants | 0 | 0

4. Primary Outcome: Safety of Ivacaftor - Number of Participants With Abnormal ECG (Prolonged QT Intervals)
Description: Number of participants with abnormal changes in their screening ECGs is another factor that will be used to evaluate the safety of ivacaftor.
Time Frame: From Screening to Day 98
Measure: Count of Participants; unit: Participants
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 29 | 10
Participants | 1 | 1

5. Secondary Outcome: Central CFTR Activity Measured by Mucociliary Clearance (MCC) Percentage Clearance at 60 Mins
Description: Clearance of Tc99 sulfur colloid is a measure of MCC of the lungs, and is calculated by a standard protocol developed by the Cystic Fibrosis Therapeutics Development Network. The method provides a robust measure of MCC, and has been sensitive to the effects of inhaled pharmacologic agents in CF and COPD including improvements of an unprecedentedly large magnitude in CF patients with the G551D-CFTR mutation treated with ivacaftor measured in a multicenter study. The technique allows estimates of MCC in both the small and large airway compartments.
Time Frame: From Screening to Day 84
Measure: Mean (Standard Deviation); unit: percentage of clearance
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 29 | 10
percentage of clearance
  Screening | 88.4 (12) | 86.2 (7)
  Day 84 | 86 (17) | 80 (2)

6. Secondary Outcome: Peripheral CFTR Activity Measured by Change in Sweat Chloride
Description: Sweat chloride abnormality is correlated with COPD severity and symptoms, and is a highly sensitive outcome measure for CFTR-directed therapeutics. We have shown sweat chloride is sensitive to the presence of cigarette smoking and COPD, and the test has been successfully used as an endpoint in multiple CF trials, including studies to detect the efficacy of ivacaftor therapy.
Time Frame: From Screening to Day 84
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 30 | 10
mmol/L | 3.9 (9.8) | 3.8 (12.1)

7. Secondary Outcome: Indicators of Respiratory Function and COPD Health : Change in FEV1 Predict %
Description: Spirometry is a standard outcome measure in COPD and a major indicator of efficacy and safety in COPD clinical trials. Post-bronchodilator spirometry will be performed by ATS criteria. FEV1 will be measured in predict percentage.
Time Frame: From Screening to Day 84
Measure: Mean (Standard Deviation); unit: predict percentage
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 29 | 10
predict percentage | 1.5 (4.7) | -0.4 (7.6)

8. Secondary Outcome: San Diego Shortness of Breath Questionnaire (SOBQ)
Description: The SOBQ is a self-reported questionnaire that assesses shortness of breath while performing a variety of activities of daily living. The Minimum Clinically Important Difference (MCID) is 5.
  The SOBQ includes 24 items, using 6-point scale with 0 = "not at all" to 5 = "maximal or unable to do because of breathlessness". The sum of SOBQ score ranges from 0 to 120, with higher score indicating more breathlessness.
Time Frame: From D1 to Day 84
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 29 | 10
units on a scale | -6.25 (26.8) | -8.6 (12.2)

9. Secondary Outcome: Breathlessness, Cough, and Sputum Scale (BCSS)
Description: The BCSS is a three-item questionnaire rating breathlessness, cough and sputum on a 5-point Likert scale from 0 (no symptoms) to 4 (severe symptoms).
  The BCSS score ranges from 0 to 12; the higher the score indicates the worse of symptoms.
Time Frame: From D1 to Day 84
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 29 | 10
units on a scale | -0.6 (2.8) | -1.2 (1.3)

10. Secondary Outcome: COPD Assessment Test (CAT)
Description: CAT is a self-reported questionnaire that measures COPD related quality of life. The MCID is 2.
  CAT composes of 8 questions, and the scores range from 0 - 40. Higher scores denote a more severe impact of COPD on a patient's life.
Time Frame: From D1 to Day 84
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 29 | 10
units on a scale | -0.7 (6.9) | -1 (6.7)

11. Secondary Outcome: St. George Respiratory Questionnaire (SGRQ)
Description: The SGRQ is a disease-specific measure of health status for use in COPD with an MCID of 4.
  The scores range from 0 to 100, with higher scores indicating more limitations.
Time Frame: From D1 to Day 84
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 29 | 10
score on a scale | -7.6 (21.0) | -10.1 (10.6)

ADVERSE EVENTS:
Time Frame: Screening to Day 98
Arm/Group | Ivacaftor | Placebo
All-Cause Mortality (participants affected / at risk) | 19/29 | 6/10
Serious Adverse Events (participants affected / at risk) | 6/29 | 1/10
Other Adverse Events (participants affected / at risk) | 0/29 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivacaftor (N=29) | Placebo (N=10)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Altered mental status (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
AECOPD (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT03085485/Prot_SAP_000.pdf